CLINICAL TRIAL: NCT03706963
Title: Remote Telemonitoring to Improve Prehabilitation and Surgical Outcomes of Patients Undergoing Elective Abdominal Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Intervention is no longer being used
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other); BJC Innovative Lab (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201810002
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Abdominal Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phone Call (Experimental): * Patients will be provided with a Fitbit wristband & assistance to set up on smart phone
  * Preoperative baseline data (activity, sleep, heartrate) will be collected for at least 14 days until the day prior to surgery
  * The group will receive a phone call 7 days into their preoperative period to identify barriers, provide available resources, & encourage continuation of prehabilitation activities
  * The physician extender will talk with the patient to identify barriers to prehabilitation activities that the patient may have experienced during the first 7 days of activity tracking & provide recommendations & resources to overcome those barriers when possible. The physician extender will encourage the patient to continue prehabilitation activities until the day of operation to meet goals. Following surgery, we will analyze Fitbit data to determine if the intervention had an impact on the patient's prehabilitation activity with the non-intervened patient group used as a control
  Interventions: Other: Phone Call
- No Phone Call (No Intervention): * Eligible patients will be provided with a Fitbit wristband & assistance to set up on smart phone
  * Preoperative baseline data (activity, sleep, heartrate) will be collected for at least 14 days until the day prior to surgery

INTERVENTIONS:
Other: Phone Call — -phone call 7 days (+/- 2 days) into preoperative period
  Arms: Phone Call

SUMMARY:
There is data confirming that simple tests of physical capability, such as the timed "get-up-and-go" test and the 6-minute walk test, correlate with surgical outcomes. It is reasonable to assume that preoperative telemonitoring, which allows for the tracking of more variables over a wider range of activities, could provide a significantly more accurate picture of a patient's physical fitness than a short one-time test performed in the clinic setting.

Almost half of the patients who are readmitted at Washington University are readmitted for less than 4 days. The readmitted patients usually present with sepsis, are treated with antibiotics and percutaneous drainage, and are discharged home relatively quickly. Earlier identification of these patients, prior to the development of sepsis, would reduce the risks to the patient and allow for outpatient management.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo elective abdominal surgery
* At least 18 years of age
* Able to understand and willing to sign an IRB-approved informed consent document

Exclusion Criteria:

* Doesn't have access to smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the study intervention during the preoperative period to increase patients compliance with prehabilitation goals as measured by average steps per day | Baseline through 30 days after surgery discharge (approximately 45 days)
Patient compliance of telemonitoring with activity trackers as measured by percentage of time the patient is wearing the device properly | Baseline through 30 days after surgery discharge (approximately 45 days)
  -The number of heart rate data points that are collected per day is used as a proxy for determining the amount of time the patient is wearing the device properly.

CONTACTS AND LOCATIONS:
Overall Officials: Chet Hammill, M.D., MCR, FACS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu